CLINICAL TRIAL: NCT05549713
Title: The Effect of Upper Blepharoplasty on Anatomical and Functional Aspects of Vision in the Early Postoperative Period
Brief Title: The Effect of Upper Blepharoplasty on Vision Quality in the Early Postoperative Period
Status: Recruiting | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Dunja Klepo, Principal investigator, Osijek University Hospital
Other Study IDs: OsijekUH-EYEDEP
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Excess Skin of Both Eyelids; Contrast Sensitivity; Tear Film Insufficiency of Both Eyes; Corneal Topography
Keywords: Corneal topography; Contrast sensitivity; Eyelid disease; Meibomian gland dysfunction; Blepharoplasty
MeSH Terms: conditions — Eyelid Diseases; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blepharoplasty group: As a single arm study, all examinees will undergo upper blepharoplasty. Data regarding corneal topography, tear film quality and contrast sensitivity will be obtained before the surgery, seven days and one month postoperatively
  Interventions: Procedure: Upper blepharoplasty

INTERVENTIONS:
Procedure: Upper blepharoplasty — Upper eyelid surgery in local anesthesia performed by removing excess skin folds and closing with sutures placed on the skin crease.

SUMMARY:
Contrast sensitivity (CS) and tear film (TF) changes are noted in late postoperative period after upper blepharoplasty (UB), while the same was rarely investigated in the early postoperative period. The reason for aforementioned improvement of vision quality is unclear. Suggested explanations include changes in higher-order aberrations, elimination of the overlay effect created by excess skin on the upper eyelids and/or eyelashes directed toward the eyelid, or changes in corneal topography (CT) and keratometry.

Furthermore, there is no consensus on the best technique for UB. Due not only to different surgical techniques, but also to different methods of measuring the tear film quality, it is very difficult to quantify the aforementioned studies.

While changes in tear volume parameters and changes in tear film (TF) rupture have been investigated in detail, changes in the lipid layer have rarely been investigated.

According to previous studies, there are different findings about changes in CT after UB.

The aim of the research is to determine whether there are anatomical (CT) and functional (TF and CS) changes in subjects with functional dermatochalasis before the procedure and in a month-long postoperative period.

The research is conducted on examinees diagnosed by clinical examination with functional dermatochalasis with the exclusion of examinees with ocular or systemic conditions affecting TF, best corrected visual acuity or CT.

Detailed medical history and ophthalmologic examination will be performed with grading of the external appearance of the upper eyelids. All diseases and conditions that can lead to changes in CS, TF or corneal defects will be noted. Preoperatively all subjects will have CS recorded in photopic conditions, TF analysis and CT (Keratograph 5M, OCULUS Optikgeraete GmbH, Wetzlar, Germany). UB will be performed in the operating room at the UED. At first (seven days postoperatively) and second (one month postoperative) check-up a CS check will be performed at the UED and TF analysis and CT at Lens LTD.

DETAILED DESCRIPTION:
Dermatochalasis is an age-related condition characterized by the development of folds of excess skin on the upper eyelid with loss of skin elasticity. The mechanical pressure created by the accumulation of excess fat tissue and skin over the upper eyelid leads to a feeling of heaviness and narrowing of the peripheral visual field, which is an indication for surgical treatment. In addition to widening the field of vision, it has been noted that upper blepharoplasty (UB) also has an impact on the subjective improvement of vision postoperatively. Although no difference in best corrected visual acuity was observed pre- and postoperatively, it was noted that contrast sensitivity (CS) improves after UB, especially in the late postoperative period, while the same was rarely investigated in the early postoperative period. The exact reason for the postoperative increase in CS is not clear. Suggested explanations include changes in higher-order aberrations, elimination of the overlay effect created by excess skin on the upper eyelids and/or eyelashes directed toward the eyelid, or changes in corneal topography (CT) and keratometry.

Furthermore, there is no consensus on the best technique for UB. Due not only to different surgical techniques, but also to different methods of measuring the tear film quality, it is very difficult to quantify the aforementioned studies.

While changes in tear volume parameters and changes in tear film (TF) rupture have been investigated in detail, changes in the lipid layer have rarely been investigated.

According to previous studies, there are different findings about changes in CT after UB.

The aim of the research is to determine whether there are anatomical (CT) and functional (TF and CS) changes in subjects with functional dermatochalasis before the procedure and in a month-long postoperative period.

The research is conducted on examinees diagnosed by clinical examination with functional dermatochalasis. Functional dermatochalasis is considered excess skin on the upper eyelid with subjective difficulties due to obstructing the upper part of visual field: swelling of the eyelids in the morning with difficulties in opening the eyes, use of the frontal musculature to be able to have at least a partial width of the field of vision in the upper part that is adequate for daily functioning, and headaches. Exclusion criteria are: history of corneal refractive surgery, pterygium, glaucoma, nuclear sclerosis > 4th degree, severe dry eye, age-related macular degeneration, neuro-ophthalmological diseases, use of hormone therapy, diabetic retinopathy or condition after panretinal photocoagulation. Corneal pathologies such as keratoconus and gross eyelid malposition conditions such as entropion, ectropion and marked laxity of the eyelids are also grounds for exclusion from the study.

The external appearance of the upper eyelids of all subjects will be graded in accordance with previous studies. All subjects will have a detailed personal and ophthalmological history taken, and a biomicroscope examination of the anterior segment and fundus. All diseases and conditions that can lead to changes in CS, TF or corneal defects will be noted. Preoperatively all subjects will have CS recorded in photopic conditions using the Pelli-Robson table, TF analysis and CT (Keratograph 5M, OCULUS Optikgeraete GmbH, Wetzlar, Germany). The CS test will be performed at the University Eye Department, University Hospital Center Osijek (UED), while the TF analysis and CT will be performed at Lens LTD, Zrinjevac 4, 31000 Osijek, completely free of charge. The need for cooperation with Lens LTD arose due to the fact that at UED there is no device for testing the function of the TF, as well as no apparatus for CT. UB will be performed in the operating room at the UED using technique of removing only excess skin without the underlying part of the orbicularis muscle from the upper eyelids. At first (seven days postoperatively) and second (one month postoperative) check-up a CS check will be performed at the UED and TF analysis and CT at Lens LTD. All data will be statistically processed and used in the form of congress announcements and scientific papers in the journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with functional dermatochalasis on the upper eyelid with subjective difficulties due to obstructing the upper part of visual field: swelling of the eyelids in the morning with difficulties in opening the eyes, use of the frontal musculature to be able to have at least a partial width of the field of vision in the upper part that is adequate for daily functioning, and headaches.

Exclusion Criteria:

* History of corneal refractive surgery, pterygium, glaucoma, nuclear sclerosis > 4th degree, severe dry eye, age-related macular degeneration, neuro-ophthalmological diseases, use of hormone therapy, diabetic retinopathy or condition after panretinal photocoagulation. Corneal pathologies such as keratoconus and gross eyelid malposition conditions such as entropion, ectropion and marked laxity of the eyelids are also grounds for exclusion from the study.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Examinees complaining of subjective difficulties due to excess skin on the upper eyelid. All examinees will be examined in University Eye Department, University Hospital Osijek
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Contrast sensitivity | Measurement will take place preoperatively, 7 days and one month postoperatively. Planned duration of the examination is five minutes
  Measurement of contrast sensitivity using Pelli-Robson chart with best corrected visual acuity in photopic condions

SECONDARY OUTCOMES:
Corneal topography | Measurement will take place preoperatively, 7 days and one month postoperatively. Planned duration of the examination is thirty minutes
  Measurement of corneal topography using Keratograph 5M, OCULUS Optikgeraete GmbH, Wetzlar, Germany
Tear film quality | Measurement will take place preoperatively, 7 days and one month postoperatively. Planned duration of the examination is thirty minutes
  Measurement of tear film quality using Keratograph 5M, OCULUS Optikgeraete GmbH, Wetzlar, Germany

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Bajtl, Principal Investigator — Osijek University Hospital
Locations (1):
- Osijek University Hospital, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeAngelis DD, Carter SR, Seiff SR. Dermatochalasis. Int Ophthalmol Clin. 2002 Spring;42(2):89-101. doi: 10.1097/00004397-200204000-00009. No abstract available. PMID 11914706
- [Background] Hacker HD, Hollsten DA. Investigation of automated perimetry in the evaluation of patients for upper lid blepharoplasty. Ophthalmic Plast Reconstr Surg. 1992;8(4):250-5. doi: 10.1097/00002341-199212000-00003. PMID 1476973
- [Background] An SH, Jin SW, Kwon YH, Ryu WY, Jeong WJ, Ahn HB. Effects of upper lid blepharoplasty on visual quality in patients with lash ptosis and dermatochalasis. Int J Ophthalmol. 2016 Sep 18;9(9):1320-4. doi: 10.18240/ijo.2016.09.15. eCollection 2016. PMID 27672599
- [Background] Nalci H, Hosal MB, Gunduz OU. Effects of Upper Eyelid Blepharoplasty on Contrast Sensitivity in Dermatochalasis Patients. Turk J Ophthalmol. 2020 Jun 27;50(3):151-155. doi: 10.4274/tjo.galenos.2019.95871. PMID 32631001
- [Background] Bhattacharjee K, Misra D, Singh M, Deori N. Long-term changes in contrast-sensitivity, corneal topography and higher-order aberrations after upper eyelid blepharoplasty: A prospective interventional study. Indian J Ophthalmol. 2020 Dec;68(12):2906-2910. doi: 10.4103/ijo.IJO_907_20. PMID 33229668
- [Background] Kiang L, Deptula P, Mazhar M, Murariu D, Parsa FD. Muscle-sparing blepharoplasty: a prospective left-right comparative study. Arch Plast Surg. 2014 Sep;41(5):576-83. doi: 10.5999/aps.2014.41.5.576. Epub 2014 Sep 15. PMID 25276652
- [Background] Zhang S, Yan Y, Lu Y, Zhou Y, Fu Y. Effect of Transcutaneous Upper Eyelid Blepharoplasty on Blink Parameters and Lipid Layer Thickness. Front Med (Lausanne). 2021 Nov 22;8:732041. doi: 10.3389/fmed.2021.732041. eCollection 2021. PMID 34881256
- [Background] Soares A, Faria-Correia F, Franqueira N, Ribeiro S. Effect of superior blepharoplasty on tear film: objective evaluation with the Keratograph 5M - a pilot study. Arq Bras Oftalmol. 2018 Nov./Dec.;81(6):471-474. doi: 10.5935/0004-2749.20180094. Epub 2018 Oct 8. PMID 30304089
- [Background] Zloto O, Matani A, Prat D, Leshno A, Ben Simon G. The Effect of a Ptosis Procedure Compared to an Upper Blepharoplasty on Dry Eye Syndrome. Am J Ophthalmol. 2020 Apr;212:1-6. doi: 10.1016/j.ajo.2019.11.021. Epub 2019 Nov 23. PMID 31770512
- [Background] Zinkernagel MS, Ebneter A, Ammann-Rauch D. Effect of upper eyelid surgery on corneal topography. Arch Ophthalmol. 2007 Dec;125(12):1610-2. doi: 10.1001/archopht.125.12.1610. PMID 18071108
- [Background] Dogan E, Akbas Kocaoglu F, Yalniz-Akkaya Z, Elbeyli A, Burcu A, Ornek F. Scheimpflug imaging in dermatochalasis patients before and after upper eyelid blepharoplasty. Semin Ophthalmol. 2015 May;30(3):193-6. doi: 10.3109/08820538.2013.839803. Epub 2014 Jan 10. PMID 24409940
- [Background] Simsek IB, Yilmaz B, Yildiz S, Artunay O. Effect of Upper Eyelid Blepharoplasty on Vision and Corneal Tomographic Changes Measured By Pentacam. Orbit. 2015;34(5):263-7. doi: 10.3109/01676830.2015.1057292. Epub 2015 Jul 17. PMID 26186387
- [Background] Shah M, Lee G, Lefebvre DR, Kronberg B, Loomis S, Brauner SC, Turalba A, Rhee DJ, Freitag SK, Pasquale LR. A cross-sectional survey of the association between bilateral topical prostaglandin analogue use and ocular adnexal features. PLoS One. 2013 May 1;8(5):e61638. doi: 10.1371/journal.pone.0061638. Print 2013. PMID 23650502